CLINICAL TRIAL: NCT05162820
Title: Impact of Solarplast® on Immunity in Active Smokers and Non-smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Deerland Probiotics and Enzymes (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2021-416
Record Dates: First submitted 2021-12-08; First posted 2021-12-17 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Immunity; Smoking, Cigarette
Keywords: Solarplast; Spinach; Skin Health
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Study
Who Masked: Participant, Investigator
Masking Description: Capsules will be of similar appearance and provided in un-identified bottles (A,B)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Smoker Solarplast (Experimental): Smoker's assigned to solarplast
  Interventions: Dietary Supplement: 100 mg Solarplast
- Smoker Placebo (Placebo Comparator): Smoker's assigned to placebo
  Interventions: Dietary Supplement: Placebo
- Non-smoker Solarplast (Experimental): Non-smoker assigned to solarplast
  Interventions: Dietary Supplement: 100 mg Solarplast
- Non-smoker Placebo (Placebo Comparator): Non-smoker assigned to placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 100 mg Solarplast — 100 mg Solarplast delivered in capsules with the carrier of rice dextrin and medium chain triglycerides consumed daily at breakfast for 60 days
  Arms: Non-smoker Solarplast; Smoker Solarplast
Dietary Supplement: Placebo — rice dextrin and medium chain triglycerides in capsules consumed daily at breakfast for 60 days
  Arms: Non-smoker Placebo; Smoker Placebo

SUMMARY:
The purpose of this study is to determine the impact of Solarplast treatment on measures of oxidative stress, immune function, skin appearance, and associated measures in 60 men and women, consisting of both cigarette smokers and nonsmokers. The hypothesis is that the Solarplast treatment will reduce oxidative stress biomarkers and favorably impact immune measures and both perceived and quantifiable measures of skin health, in both smokers and non-smokers, with a greater impact observed in smokers. Photographic analyses like the Pear Plus 3D system have been developed for clinical use for monitoring skin health.

DETAILED DESCRIPTION:
Deerland Probiotics and Enzymes has developed a dietary supplement called Solarplast®, which is an organic spinach extract, currently being sold on the market (Solarplast - Deerland Probiotics and Enzymes). It contains a unique mixture of antioxidant enzymes and single antioxidant molecules that work to attack reactive oxygen species (ROS) through chaperone activity. These chaperones are naturally occurring proteins that provide protection from stress, such as ROS, heat, and infection, and can lead to reduced inflammation and alteration in immune function.

Spinach is rich in select vitamins and minerals, such as iron, vitamin A, riboflavin, and lutein-a carotenoid that acts as a natural antioxidant, protecting the body from toxins and ROS. Solarplast is thought to exhibit antioxidant protection against ROS, while also containing photosynthetic complexes with high concentrations of ATP, NADPH, ADP, AMP, NADP, niacin, B12, adenine, and ribose. Therefore, it may provide the components required to scavenge free radicals and mitigate ensuing damage from ROS.

In living cells, ROS such as singlet oxygen (·O), superoxide radical (O2· -), and hydroxyl radical (·OH) are continuously formed as a consequence of normal cellular metabolism and are increased under conditions of environmental stress. Production of ROS in quantities that overwhelm the endogenous antioxidant defense system leads to oxidative stress, and this oxidative stress is strongly linked to the pathogenesis of numerous diseases, including diabetes, cancer, and cardiovascular disease.

Oxidative stress leads to increases in proinflammatory cytokines such as IL-1B and TNF-alpha. Lipopolysaccharide (LPS) can induce ROS and proinflammatory cytokines. Antioxidants present in spinach may provide some protection against LPS actions.

It is well known that cigarette smoking exacerbates ROS formation and poses a significant pro-oxidant stress in vivo. In one puff of a cigarette, the smoker is exposed to >1015 free radicals in the gas phase alone, with additional exposure in the tar phase equal to >1017 free radicals·g-1. This direct exposure represents only a fraction of the total oxidative stress experienced, as cigarette smoke contributes to further endogenous ROS production mediated through inflammatory and immune processes. ROS formation due to cigarette smoking is thought to contribute to premature skin aging . Carotenoids like lutein in spinach, are believed to help protect skin from this ROS damage. Therefore, treating smokers with antioxidant therapy may not only alter immune function and measures of oxidative stress, but also prove helpful to both perceptions and measures of skin health.

Antioxidant supplementation can also reduce oxidative stress, which is linked to cognitive/mental health. Those who are exposed to high levels of oxidants and who are in a chronic state of oxidative stress (e.g., smokers) may be more susceptible to impaired mental health.

A previous clinical research trial evaluating Solarplast titled "Efficacy of Solarplast for Health and Oxidative Stress, A Randomized, Double-Blind, Placebo-Controlled Study" noted improved antioxidant defense and immunity, as well as improved subjective feelings of health (e.g., decreased irritability, decreased tension and anxiety), and improved self-reported skin health in a sample of smokers and non-smokers. The present study seeks to extend these findings in a larger sample of smokers.

The purpose of this study is to determine the impact of Solarplast treatment on measures of oxidative stress, immune function, skin appearance, and associated measures in 60 men and women, consisting of both cigarette smokers and nonsmokers. We hypothesize that the Solarplast treatment will reduce oxidative stress biomarkers and favorably impact immune measures and both perceived and quantifiable measures of skin health, in both smokers and non-smokers, with a greater impact observed in smokers. Smoking, causes a decrease in blood flow to skin and dryness along with other adverse effects that can prematurely age skin. As quantifiable measures provide more sound evidence than personal perceptions when evaluating skin treatments, there has been a greater push for more analytical methods in the assessment of skin regimens which include topographical, pigmentation, color, as well as other measures that will be employed in this study via photographical image analysis of subject's facial skin. Photographic analyses like the Pear Plus 3D system have been developed for clinical use for monitoring skin health.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18-40 kg/m2 (not morbidly obese)
* if a smoker, smokes at least 5 cigarettes per day for the past 12 months
* if a smoker, experience occasional mild skin irritations (e.g., rash, dryness, redness, itching, etc.)
* if non-smoker, not have used tobacco products or any smoked product (e.g., marijuana, cigar, pipe) in the past 12 months
* if non-smoker, not exposed to regular second-hand smoke (e.g., lives with or works in close proximity to a smoker)
* no consumption of alcohol-containing beverages within 48 hours of testing
* no consumption of caffeine-containing beverages within 24 hours of testing
* without active infection or illness of any kind
* if female, not be pregnant
* able to fast overnight (10-12 hours)
* Not have doctor prescribed immune function or antioxidant nutritional supplements, over the counter medications, or prescription drugs that might impact outcomes (e.g. Vitamin-C, elderberry, ginger, turmeric, quercetin, supplements with "Immun" or have immunity on their label, Immunosuppressives: prednisolone, Azathioprine, Mycophenolate mofetil, Monoclonal antibodies - of which there are many ending in "mab", such as bevacizumab, rituximab and trastuzumab, Anti-TNF drugs such as etanercept, infliximab, adalimumab, certolizumab and golimumab, Methotrexate, Ciclosporin, Tacrolimus, Sirolimus, Cyclophosphamide, Leflunomide, Immunotherapies: Immune Checkpoint Inhibitors, Adoptive Cell Therapies, Monoclonal Antibodies, Oncolytic Virus Therapy, Immune System Modulators, etc.)
* be willing to stop non-prescribed immune function or antioxidant nutritional supplements and over the counter medications (e.g. Vitamin-C, elderberry, ginger, turmeric, quercetin, supplements with "Immun" or have immunity on their label, etc.) one month prior to and through the duration of the study

Exclusion Criteria:

-

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Plasma Cytokine Panel | baseline
  Cytokines analyzed from plasma for IL-1beta, IL-6, IL-10, and TNF-alpha
Plasma Cytokine Panel | after 30 days of treatment
  Plasma analyzed for IL-1beta, IL-6, IL-10, and TNF-alpha
Plasma Cytokine Panel | after 60 days of treatment
  Plasama analyzed for IL-1beta, IL-6, IL-10, and TNF-alpha
Plasma Cytokine Panel on LPS treated whole blood | baseline
  LPS treated whole blood analyzed for IL-1beta, IL-6, IL-10, and TNF-alpha
Plasma Cytokine Panel on LPS treated whole blood | after 30 days of treatment
  LPS treated whole blood analyzed for IL-1beta, IL-6, IL-10, and TNF-alpha
Plasma Cytokine Panel on LPS treated whole blood | after 60 days of treatment
  LPS treated whole blood analyzed for IL-1beta, IL-6, IL-10, and TNF-alpha
Protein oxidation | baseline
  Blood sample analyzed for protein oxidation
Protein oxidation | after 30 days of treatment
  Blood sample analyzed for protein oxidation
Protein oxidation | after 60 days of treatment
  Blood sample analyzed for protein oxidation
Lipid peroxidation | baseline
  Blood sample analyzed for lipid peroxidation
Lipid peroxidation | after 30 days of treatment
  Blood sample analyzed for lipid peroxidation
Lipid peroxidation | after 60 days of treatment
  Blood sample analyzed for lipid peroxidation
Subjects' perceived mental health | baseline
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 1 week of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 2 weeks of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 3 weeks of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 4 weeks of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 5 weeks of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 6 weeks of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 7 weeks of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subjects' perceived mental health | 8 weeks of treatment
  Subject's self-report different measures of mental health using a questionnaire with a scale of 1 (None of the time) to 5 (All of the time)
Subject's perceived general health and well-being | baseline
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 1 week of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 2 weeks of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 3 weeks of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 4 weeks of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 5 weeks of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 6 weeks of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 7 weeks of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived general health and well-being | 8 weeks of treatment
  ubject's self-report different aspects of general health and well-being using a questionnaire with a scale of 1 (None) to 5 (Severe)
Subject's perceived skin health | baseline
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 1 week of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 2 weeks of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 3 weeks of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 4 weeks of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 5 weeks of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 6 weeks of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 7 weeks of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Subject's perceived skin health | 8 weeks of treatment
  ubject's self-report their perception of their skin health for different skin qualities using a questionnaire with a scale of 1 (Very Bad) to 5 (Very Good)
Quantitative Skin measures | baseline
  A skin report will generated using the 3D Pear Plus system
Quantitative Skin measures | 30 days of treatment
  A skin report will generated using the 3D Pear Plus system
Quantitative Skin measures | 60 days of treatment
  A skin report will generated using the 3D Pear Plus system

SECONDARY OUTCOMES:
Food Logs | baseline
  Dietary intake will be reported for the 5 days prior to the study visit
Food Logs | 30 days of treatment
  Dietary intake will be reported for the 5 days prior to the study visit
Food Logs | 60 days of treatment
  Dietary intake will be reported for the 5 days prior to the study visit
Resting blood pressure | baseline
  Blood pressure will be measured following a 10 minute rest
Resting blood pressure | 30 days of treatment
  Blood pressure will be measured following a 10 minute rest
Resting blood pressure | 60 days of treatment
  Blood pressure will be measured following a 10 minute rest

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No